CLINICAL TRIAL: NCT05257369
Title: Clinical Efficacy of LED Phototherapy Devices With Blue - Green Versus Blue Light of Equal Irradiance in Neonates With Non Hemolytic Jaundice
Brief Title: Broad Band Emission LED Phototherapy Source Versus Narrow Band
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erebouni Medical Center (Other)
Responsible Party: Principal Investigator, Pavel Mazmanyan, Prof. Pavel Mazmanyan, Erebouni Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 003PH
Record Dates: First submitted 2022-02-08; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Neonatal Hyperbilirubinemia; Jaundice, Neonatal
Keywords: Phototherapy; Blue light LED; Green Light LED
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Jaundice, Neonatal

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1.Blue-Green LED wide band phototherapy (Experimental): For experimental group was used "Malysh" phototherapeutic device (Luzar ltd, Belarus); it includes of eighteen blue- green super bright LEDs (12 blue (λmax 476 ) and 6 green (505 nm).
  Interventions: Device: Blue-Green LED photoherapy
- 2.Blue LED narrow band phototherapy (Active Comparator): For control group was used blue LED BILI-THERAPY (Atom Medical Inc., Tokyo, Japan) in high-mode which have a 20 μW/cm2 with peak wavelength between (λmax 480 nm).
  Interventions: Device: Blue-Green LED photoherapy

INTERVENTIONS:
Device: Blue-Green LED photoherapy — Continuous phototherapy for 24 h, for newborns placed incubators or radiant warmers will interrupted only for feeding and nursing for 20 - 30 min every three hours.
  Other Names: Blue LED phototherapy

SUMMARY:
Phototherapy is the most frequently used treatment in neonatology when serum bilirubin levels exceed physiological limits. Light-emitting diodes (LEDs) are become routinely used for phototherapy in neonates with hyperbilirubinemia. Blue LED light with peak emission around 460 nm is regarded as the most suitable light sources for phototherapy and they recommended by most neonatal guidelines. However, the effectiveness of phototherapy with narrow-band LED light sources can be increased by expanding the spectral range of incident radiation within the absorption of bilirubin due to the strongly marked heterogeneity absorption properties of bilirubin in a different microenvironment. Longer wavelength light, such as green light, is expected to penetrate the infant's skin deeper. It is still controversial whether the use of green light has any advantage over blue light. The most effective and safest light source and the optimal method to evaluate phototherapy, however, remain unknown.The aim of this study was to compare, at equal light irradiance, the clinical efficacy of broad spectrum blue- green LED with blue narrow spectral band phototherapy device.

ELIGIBILITY:
Inclusion Criteria:

* non-haemolytic hyperbilirubinaemia, but otherwise healthy, indications for phototherapy based on NICE criteria, gestational age ≥33 weeks, birth weight ≥1800 g, postnatal age >24 hrs and ≤14 days

Exclusion Criteria:

* hemolytic jaundice, major congenital animalities and history of phototherapy. Infants with indication of intensive treatment double phototherapy were not included.

Ages: 24 Hours to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Bilirubin level reduction | 24 hours
  Reduction in TSB levels after phototherapy for 24 hours

SECONDARY OUTCOMES:
Days of phototherapy | "Through study completion, an average of 1 month.
  Duration of phototherapy

OTHER OUTCOMES:
Adverse outcomes | "Through study completion, an average of 1 month.
  Any adverse effects or patologycal symptoms during phototherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Erebouni Medical Centre, NICU, Yerevan, Armenia